CLINICAL TRIAL: NCT05728710
Title: Outcomes of Perforation After Colorectal Endoscopic Submucosal Dissection
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Marion SCHAEFER, MD, Central Hospital, Nancy, France
Other Study IDs: 2022PI178
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Colorectal Neoplasms; Perforation of Rectum; Perforation Colon
Keywords: endoscopic submucosal dissection; laterally spreading tumors; perforation
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 48 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Perforation: all patients with immediate or delayed perforation identified from the FECCO (NCT04592003)
  Interventions: Procedure: Endoscopic submucosal dissection

INTERVENTIONS:
Procedure: Endoscopic submucosal dissection — standard ESD performed and complicated with a perprocedural or delayed perforation

SUMMARY:
Endoscopic resection of superficial colorectal neoplasms decrease risk of colorectal cancer. En bloc resection is necessary for large superficial lesions with risk of superficial submucosal cancer and is advised if feasible for all lesions. Endoscopic submucosal dissection (ESD) allows en bloc resection of large superficial colorectal neoplasms, increasing curative resection rate and decreasing local recurrence risk. However, the risk of perprocedural or delayed perforation is higher compared to wild field piece meal endoscopic mucosal resection. Endoscoping clipping and closing methods mostly allow conservative treatment, but some case still necessitate surgery. The aim of our study is to describe and ananalyse outcomes after perprocedural or delayed perforation in all patients undergoing ESD and analyse the need for surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

* patients from the FECCO (NCT04592003) cohort experiencing perprocedural or delayed perforation
* age over 18 years old

Exclusion Criteria:

* patients refusing exploitations of health datas
* patient treated with endoscopic mucosal resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all adults patients identified from the FECCO (NCT04592003) cohort experciencing perprocedural or delayed perforation
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Surgery | 30 days
  Rate of surgery following perforation after ESD

SECONDARY OUTCOMES:
Hospital stay | 60 days
  length of hospital stay (days)
Hospital readmission | 30 days
Curative resection rate | 60 days
Endoscopically closed perforation rate | 30 days
Risk factors for endoscopic closure failure | 30 days
30-days mortality rate | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Marion Schaefer, MD, Principal Investigator — Central Hospital, Nancy, France
Locations (13):
- Clinique CHC, Liège, Belgium
- France (12):
  - Clinique Anjou, Angers
  - CHU Bordeaux, Bordeaux
  - CHU Dijon, Dijon
  - CHU Dupuytren, Limoges
  - Hopital Edouard Herriot, Lyon
  - Hopital Privé Jean Mermoz, Lyon
  - Nancy Hospital Center, Nancy
  - Clinique Jules Verne, Nantes
  - Hopital Europeen Georges Pompidou, Paris
  - Hôpital Cochin, Paris
  - Hôpital Saint Joseph, Paris
  - CHU de Rennes, Rennes

IPD SHARING:
Plan to Share IPD: No